CLINICAL TRIAL: NCT00343200
Title: A Multicenter, Randomized, Parallel-Group, Double-Blind, Placebo-Controlled Flexible-Dose Study To Assess The Efficacy And Safety Of Viagra (Sildenafil Citrate) In Men With Erectile Dysfunction (ED) Who Do Not Self Identify.
Brief Title: A Study Of The Safety and Efficacy Of Viagra In Men With Erectile Dysfunction Who Do Not Self Identify.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A1481247
Record Dates: First submitted 2006-06-20; First posted 2006-06-22 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Sildenafil (Experimental)
  Interventions: Drug: Viagra (sildenafil citrate)

INTERVENTIONS:
Drug: Placebo — Placebo tablet orally approximately 1 hour before sexual activity, with no more than 1 dose in a 24-hour period, for a total of 8 weeks (DB phase). In 4-week OL phase, subjects received sildenafil 50 mg or 100mg orally approximately 1 hour before sexual activity, with no more than 1 dose in a 24-hour period.
  Arms: Placebo
Drug: Viagra (sildenafil citrate) — Sildenafil 50 mg or 100mg orally approximately 1 hour before sexual activity, with no more than 1 dose in a 24-hour period, for a total of 12 weeks (8-week DB phase and 4-week OL phase).
  Arms: Sildenafil

SUMMARY:
To compare the efficacy and safety of Viagra (sildenafil citrate) vs. placebo for the treatment of men with ED and at least 1 prespecified risk factor who do not self identify as having ED.

ELIGIBILITY:
Inclusion Criteria:

* Men who do not identify as having ED with documented ED
* Men 30 years of age and older
* At least one prespecified risk factor for ED

Exclusion Criteria:

* Subjects currently prescribed, taking and/or likely to be treated with nitrates or nitric oxide donors in any form on either a regular or intermittent basis
* Subjects with a known history of retinitis pigmentosa.

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2006-07; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To determine the change from baseline in Erectile Function (EF) domain of International Index of Erectile Function (IIEF). | Week 8

SECONDARY OUTCOMES:
Other questionnaires and variables such as IIEF, SEAR, GEAQ, SEX-Q, QEQ, EDITS, SEP, Event Log, Erection Hardness Grading Score, and Morisky Compliance. | Weeks 8 and 12
Safety and Tolerability | up to 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (45):
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Rosa, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Avon, Connecticut
  - Pfizer Investigational Site, Manchester, Connecticut
  - Pfizer Investigational Site, Wilmington, Delaware
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Arkansas City, Kansas
  - Pfizer Investigational Site, Newton, Kansas
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Livonia, Michigan
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Binghamton, New York
  - Pfizer Investigational Site, Endwell, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Mogadore, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Simpsonville, South Carolina
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Oregon, Wisconsin

REFERENCES:
- [Derived] Cappelleri JC, Chambers R. Addressing Bias in Responder Analysis of Patient-Reported Outcomes. Ther Innov Regul Sci. 2021 Sep;55(5):989-1000. doi: 10.1007/s43441-021-00298-5. Epub 2021 May 27. PMID 34046875
- [Derived] Kaminetsky JC, Stecher V, Tseng LJ. Quality of erections by age group in men with erectile dysfunction. Int J Clin Pract. 2017 Oct;71(10). doi: 10.1111/ijcp.12976. Epub 2017 Sep 11. PMID 28892218
- [Derived] Shabsigh R, Kaufman J, Magee M, Creanga D, Russell D, Budhwani M. Lack of awareness of erectile dysfunction in many men with risk factors for erectile dysfunction. BMC Urol. 2010 Nov 5;10:18. doi: 10.1186/1471-2490-10-18. PMID 21054874
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481247&StudyName=A%20Study%20Of%20The%20Safety%20and%20Efficacy%20Of%20Viagra%20In%20Men%20With%20Erectile%20Dysfunction%20Who%20Do%20Not%20Self%20Identify.